CLINICAL TRIAL: NCT04495036
Title: Acceptance of Telemedicine in Dermatology Patients, Physicians and Medical Staff
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: Req-2019-00523; sp20Maul2
Record Dates: First submitted 2020-07-28; First posted 2020-07-31 (Actual); Last update posted 2020-08-04 (Actual); Status verified 2020-08

CONDITIONS: Dermatologic Disease
Keywords: Teledermatology; Telemedicine
MeSH Terms: conditions — Skin Diseases | interventions — Data Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- dermatology patients
  Interventions: Other: data collection (21-items-patient descriptive survey)
- physicians and medical staff
  Interventions: Other: data collection (23-items-physician descriptive survey)

INTERVENTIONS:
Other: data collection (21-items-patient descriptive survey) — Dermatology patients are asked to complete a 21-items-survey while waiting for the doctor's consultation. Following variables will be addressed:
  * Demographic data of telemedicine users and non-users
  * Subjective disease perception of the dermatology patients
  * Use of internet, telemedicine and telemedicine insurance model
  * Patients´ willingness for additional features of telemedicine
  * Advantages and disadvantages telemedicine and face-to-face consultation
  * Suitable fields of dermatology for telemedicine from the patient's perspective
  * Recommended structure of telemedical services by users and non-users
  Groups: dermatology patients
Other: data collection (23-items-physician descriptive survey) — To obtain the view of Swiss dermatologists, other physicians and medical staff on telemedicine a 23-items-survey will be completed. Following variables will be addressed:
  * Objective disease perception of the treating dermatologist (regarding the urgency of the patient's medical examination, the functional impairment and cosmetic burden due to patient's disease, the impairment of life quality due to patient's disease and the estimation of the course of the patient's disease)
  * Suitable fields of dermatology for telemedicine from the physician's and medical staff's perspective
  Groups: physicians and medical staff

SUMMARY:
This study is to investigate the current use and intention to use of teledermatology in Swiss dermatology patients, dermatologists, other physicians and medical staff.

DETAILED DESCRIPTION:
Telemedicine, the use of telecommunication and information technology to provide clinical health care from a distance, has become an increasing role in basic medical care internationally. Telemedicine is particularly suitable for skin diseases. In order to improve the use of evidence-based telemedicine, the Swiss patients' preferences regarding teledermatology versus face-to-face consultations and the patients' and physicians' determinants of acceptance for teledermatology are investigated in this study. Dermatology patients are asked to complete a newly-created 21-items-survey; Swiss dermatologists, other physicians and medical staff on telemedicine will complete a similar newly-created, 23-items-questionnaire. A descriptive statistical analysis (e.g. gender, age, place of residence (city or country), waiting time) will be performed.

ELIGIBILITY:
Inclusion Criteria:

* patients treated in the Department of Dermatology of the Cantonal Hospital Aarau and the University Hospitals Basel and Zürich
* dermatologists, other physicians and medical staff of the Department of Dermatology of the Cantonal Hospital Aarau and the University Hospitals Basel and Zürich

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients treated in the Department of Dermatology of the Cantonal Hospital Aarau and the University Hospitals Basel and Zürich and Dermatologists, other physicians and medical staff of the Department of Dermatology of the Cantonal Hospital Aarau and the University Hospitals Basel and Zürich.
Sampling Method: Probability Sample
Enrollment: 683 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2020-01-31 (Actual); Study Completion 2020-01-31 (Actual)

PRIMARY OUTCOMES:
descriptive analysis: deviation in influencing factors for the acceptance of teledermatology | at baseline
  Assessment of the deviation in influencing factors for the acceptance of teledermatology (subjective disease perception versus objective assessment by physicians)
descriptive analysis of the impact of medical education for the acceptance of telemedicine among dermatologists vs. other physicians vs. medical staff vs. patients | at baseline
  Comparison of the impact of medical education for the acceptance of telemedicine among dermatologists vs. other physicians vs. medical staff vs. patients

CONTACTS AND LOCATIONS:
Overall Officials: Lara Valeska Maul, Dr. med., Principal Investigator — Department of Dermatology, University Hospital Basel
Locations (3):
- Switzerland (3):
  - Kantonsspital Aarau, Aarau
  - Department of Dermatology, University Hospital Basel, Basel
  - University Hospital Zürich, Zurich

REFERENCES:
- [Derived] Maul LV, Jahn AS, Pamplona GSP, Streit M, Gantenbein L, Muller S, Nielsen ML, Greis C, Navarini AA, Maul JT. Acceptance of Telemedicine Compared to In-Person Consultation From the Providers' and Users' Perspectives: Multicenter, Cross-Sectional Study in Dermatology. JMIR Dermatol. 2023 Aug 11;6:e45384. doi: 10.2196/45384. PMID 37582265